CLINICAL TRIAL: NCT05960487
Title: Can Multifidus Muscle Area Affect Cervical Interlaminar Epidural Steroid Injection Outcomes?
Brief Title: Effect of Cervical Multifidus Muscle Area on Interlaminar Epidural Steroid Injection Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.1203
Record Dates: First submitted 2023-07-09; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The patients with a significant decrease in pain severity: Evaluation will be done separately in the 3rd week and 3rd month follow-up periods of the cervical epidural steroid injection. Numerical rating scale (NRS) will be used to evaluate pain severity. A reduction of at least 50 percent in the NRS score will be considered significant.
  Interventions: Other: Cervical multifidus muscle area measurement at 3 levels (C4-C5, C5-C6, C6-C7)
- Patients without significant decrease in pain severity: Evaluation will be done separately in the 3rd week and 3rd month follow-up periods of the cervical epidural steroid injection. Numerical rating scale (NRS) will be used to evaluate pain severity. A reduction of at least 50 percent in the NRS score will be considered significant.
  Interventions: Other: Cervical multifidus muscle area measurement at 3 levels (C4-C5, C5-C6, C6-C7)

INTERVENTIONS:
Other: Cervical multifidus muscle area measurement at 3 levels (C4-C5, C5-C6, C6-C7) — Cervical multifidus muscle area measurement will be performed from both the side affected by radiculopathy and the unaffected side using the magnetic resonance (MR) imaging. Measurements will be made by two researchers, independent of each other.

SUMMARY:
Cervical radiculopathy is one of the most important causes of chronic neck pain. Cervical epidural steroid injections including interlaminar approach are frequently used for treatment option in patients that more conservative modalities are ineffective.

Paraspinal muscles have an important role in supporting neck movements and providing stability of the cervical spine. The multifidus muscle, located in the deepest part of the neck extensor muscle group, has become the muscle that is frequently emphasized in spinal pain in recent years. In the literature, it has been shown that the multifidus muscle on the affected side is atrophied in patients with cervical radiculopathy.

Although many factors are known to be effective on the outcomes of cervical interlaminar epidural injection, there are limited data on the effect of the multifidus muscle area. In this retrospective study, it was planned to investigate the effect of the multifidus muscle area on the results of cervical interlaminar epidural steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral radicular pain due to cervical disc herniation for at least 3 months
* Patients with disc herniation level C5-C6
* Patients who are unresponsive to other conservative treatments and who have undergone cervical interlaminar epidural steroid injection

Exclusion Criteria:

* Patients with incomplete medical records (absence of MR imaging, incomplete data of 3rd week and 3rd month follow-up periods after cervical interlaminar epidural steroid injection)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have cervical disc herniation at the C5-C6 level and have radicular pain complaints for at least 3 months will be included in the study. Cervical interlaminar epidural steroid injection was applied to the patients and their follow-ups at the 3rd week and 3rd month should have been recorded completely.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-07 (Estimated)

PRIMARY OUTCOMES:
Cervical multifidus muscle area | Through study completion, an average of 2 weeks
  Multifidus muscle measurement will be performed at 3 levels (C4-C5, C5-C6, C6-C7) in the MR imaging obtained from the medical records of the participants in both groups and the values will be compared with each other. Difference between muscle areas will be evaluated for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Gunay Yolcu, M.D., Principal Investigator — Marmara University; Osman Hakan Gunduz, Prof., Study Chair — Marmara University

IPD SHARING:
Plan to Share IPD: Undecided